CLINICAL TRIAL: NCT05294718
Title: External Shunt Versus Internal Shunt for Off Pump Glenn (Original Article)
Brief Title: : External Shunt Versus Internal Shunt for Off Pump Glenn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Elhaddad, Lecturer of Anesthesia, ICU and Pain managment, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-103-2013
Record Dates: First submitted 2022-02-26; First posted 2022-03-24 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Intervention Model Description: A prospective, randomized comparative study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: concealed in opaque closed envelops
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal shunt (Active Comparator): glenn with internal shunt (veno-atrial shunt) where the surgeon established a shunt between distal SVC and the right atrium, Establishing a veno-atrial shunt.
  Interventions: Procedure: Internal shunt
- External shunt (Active Comparator): Glenn with external shunt where the anesthesiologist connected the internal Jagular venous cannula which represent the SVC with the main lumen of the femoral cannula which represent the IVC through long venous extension
  Interventions: Procedure: External shunt

INTERVENTIONS:
Procedure: Internal shunt — glenn with internal shunt (veno-atrial shunt) where the surgeon established a shunt between distal SVC and the right atrium, Establishing a veno-atrial shunt.
  Other Names: Venoatrial shunt
  Arms: Internal shunt
Procedure: External shunt — Glenn with external shunt where the anesthesiologist connected the internal Jagular venous cannula which represent the SVC with the main lumen of the femoral cannula which represent the IVC through long venous extension
  Other Names: Jagulo femoral shunt
  Arms: External shunt

SUMMARY:
A prospective, randomized comparative study where investigators present results of off pump bidirectional Glenn operation done using either a venoatrial shunt or external shunt to decompress superior vena cava during clamping.

DETAILED DESCRIPTION:
The bidirectional Glenn shunt (BDG) is performed for cyanotic congenital heart defects, with single-ventricle pathology . The BDG is usually performed with cardiopulmonary bypass (CPB) with its associated complications. The conduct of this operation without CPB can be associated with elevation of superior vena caval (SVC) pressure that may lead to neurological damage.

However, the safety of performing BDG without CPB reported by many authors but with some decompression techniques of the SVC at the time of clamping

Objective: investigators present results of off pump bidirectional Glenn operation done using either a venoatrial shunt or external shunt to decompress superior vena cava during clamping.

Design A prospective, randomized comparative study Setting: Single tertiary care cardiac center Participants 30 patients with functional single ventricle who will go off pump bidirectional Glenn.

Interventions: The patients will be randomly assigned into two groups: Group I (n = 15), where it will be done with a veno-atrial shunt(internal), and Group II (n = 15), where it will be done with an external shunt. All patients will go a complete neurological examination both preoperatively as well as postoperatively Intraoperative data will be collected and analyzed at the following time points: pre-clamping (post induction), during clamping and after de-clamping of SVC. variables such as arterial oxygen saturation (SaO2), systolic blood pressure (SBP), mean arterial blood pressure (MAP), diastolic blood pressure (DBP), and hematocrit, CVP, SVC pressure, cerebral perfusion pressure (CPP= MAP-CVP), PaO2, PaCO2 and ScvO2 will be analyzed.

Postoperatively, the patients will be stabilized in the intensive care unit (ICU) and after monitoring the SVC pressure for 12 h, the internal jugular vein cannula will be removed to prevent any jugular vein thrombosis. The patients will start aspirin (5 mg/kg/day), which will be continued indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* single-ventricle lesions,
* good sized branch pulmonary arteries (Magoon's index > 1.5),
* PA pressures < 20 mmHg,
* So2 < 80%,
* age range from (6 months-5years)
* weight range from (6-21) kg, -All these patients had adequate atrial septal defects and none of these patients required any intra cardiac repair.-

Exclusion Criteria:

* previous cardiac operation,
* known intracranial pathology,
* neurologic disease
* craniofacial anomalies.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Mean SVC Pressure | during SVC clamping procedure
  Measurment of superior vena cava pressure during off pumb Glenn

SECONDARY OUTCOMES:
mean ABP | "baseline, pre-intervention" "during the intervention procedure" "immediately after the intervention
  Measurment of mean arterial blood preassure during off bumb Glenn
cerebral perfusion pressure | "baseline, pre-intervention" "during the intervention procedure" "immediately after the intervention
  CPP= MABP - CVP
Mean SVC clamp time | during SVC clamping procedure
  Duration of SVC during off pump glenn with either Internal or external shunt

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy hospital, Cairo, Egypt